CLINICAL TRIAL: NCT02038920
Title: Phase III, Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Intravenous MLN0002 (300 mg) Infusion in Induction and Maintenance Therapy in Japanese Subjects With Moderate or Severe Crohn's Disease
Brief Title: Phase III Study of MLN0002 (300 mg) in Treatment of Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN0002/CCT-001; U1111-1150-2688 (Other: WHO); JapicCTI-142402 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Induction Phase: Vedolizumab, 300 mg (Experimental): Vedolizumab 300 mg, intravenous (IV) infusion, once at Weeks 0, 2 and 6 in the induction phase.
  Interventions: Drug: Vedolizumab
- Induction Phase: Placebo (Placebo Comparator): Vedolizumab placebo-matching IV infusion once at Weeks 0, 2 and 6 in the induction phase.
  Interventions: Drug: Vedolizumab placebo
- Maintenance Phase: Vedolizumab 300 mg (Experimental): Vedolizumab placebo-matching, IV infusion, once at Weeks 14, 22, 30, 38, 46 and 54 in maintenance phase. Participants received vedolizumab in induction phase and achieved Crohn's Disease Activity Index (CDAI)-70 response at Week 10 and were randomized to receive vedolizumab in maintenance phase.
  Interventions: Drug: Vedolizumab
- Maintenance Phase: Placebo (Placebo Comparator): Vedolizumab placebo-matching, IV infusion, once at Weeks 14, 22, 30, 38, 46 and 54 in maintenance phase. Participants received vedolizumab in induction phase and achieved CDAI-70 response at Week 10 and were randomized to receive placebo in maintenance phase.
  Interventions: Drug: Vedolizumab placebo
- Maintenance Phase: Placebo Continuation (Placebo Comparator): Vedolizumab placebo-matching, IV infusion, once at Weeks 14, 22, 30, 38, 46 and 54 in maintenance phase. Participants received vedolizumab placebo-matching in induction phase and achieved CDAI-70 response at Week 10 received placebo in maintenance phase without randomization.
  Interventions: Drug: Vedolizumab placebo
- Open-Label: Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once at Weeks 0, 2 and 6 and then every 8 weeks thereafter up to Week 94 as a maximum duration in open-label phase.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV injection
  Other Names: MLN0002
  Arms: Induction Phase: Vedolizumab, 300 mg; Maintenance Phase: Vedolizumab 300 mg; Open-Label: Vedolizumab 300 mg
Drug: Vedolizumab placebo — Vedolizumab placebo-matching IV infusion
  Arms: Induction Phase: Placebo; Maintenance Phase: Placebo; Maintenance Phase: Placebo Continuation

SUMMARY:
This study is a phase 3, multicenter, randomized, double-blinded, placebo-controlled, parallel-group study to examine the efficacy, safety, and pharmacokinetics of vedolizumab (MLN0002) in induction and maintenance therapy in Japanese participants with moderately or severely active Crohn's disease.

DETAILED DESCRIPTION:
This is a phase 3, multicenter, randomized, double-blinded, placebo-controlled, parallel-group study to examine the efficacy, safety, and pharmacokinetics of intravenous vedolizumab (300 mg) infusion in induction and maintenance therapy in Japanese participants with moderately or severely active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, participants were capable of understanding and complying with protocol requirements
2. Participants or, when applicable, participants legally acceptable representative sign and date the informed consent form prior to initiation of any study procedures
3. Participants aged 15 to 80 years (inclusive) at the time of consent
4. A nonsterilized male participant who has a female partner of child-bearing potential has to agree to use adequate contraception during the period from the signing of informed consent to 6 months after the last dose of the study drug
5. A female participant of child-bearing potential (i.e., nonsterilized or whose last regular menses was within previous 2 years) who has a nonsterilized male partner has to agree to use adequate contraception during the period from the signing of informed consent to 6 months after the last dose of the study drug
6. Participants with a diagnosis of small-intestinal, large-intestinal, or small-/large-intestinal Crohn's disease (CD) established based on the Revised Diagnostic Criteria for Crohn's disease issued by Research Group for Intractable Inflammatory Bowel Disease Designated as Specified Disease by the Ministry of Health, Labor and Welfare of Japan (2012) at least 3 months before the start of administration of study drug
7. Participants with baseline CDAI score of 220 to 450(inclusive) and meeting at least one of the followings:

   * C-reactive protein (CRP) at screening test is above 0.30 mg/dL
   * Participants with irregular or semicircular ulcers or multiple aphthae (10 or more) observed over an extensive area of the small or large intestine on endoscopy or imaging test within the 4 months before the start of administration of study drugs
   * Participants with longitudinal ulcers or a cobblestone appearance observed in the small or large intestine on endoscopy or imaging test within 4 months before the start of administration of study drugs
8. In case of the participants who meet any of the following criteria; participants with ≥ 8-year history of extensive or limited colitis, participants aged ≥ 50 years, or participants with a first-degree family history of colon cancer, those whom the complication of colon cancer or dysplasia was ruled out by total colonoscopy at the start of study drug administration (or the results from total colonoscopy performed within 1 year before giving consent are available)
9. Participants meeting the criteria for treatment failure below with at least one of the following agents received within previous 5 year period before giving consent

   1. Corticosteroids

      * Resistance
      * Dependence
      * Intolerance
   2. Immunomodulators (azathioprine, 6-mercaptopurine or methotrexate)

      * Refractory
      * Intolerance
   3. Anti-tumor necrosis factor alpha (TNFα) antibodies

      * Inadequate response
      * Loss of response
      * Intolerance

Exclusion Criteria:

1. Participants with an evidence of or suspected abdominal abscess
2. Participants with a history of subtotal or total colectomy
3. Participants who have had a resection of the small intestine in at least 3 locations or have a diagnosis of short bowel syndrome
4. Participants with ileostomy, colostomy, or internal fistula, or severe intestinal stenosis
5. Participants who have a treatment history with natalizumab, efalizumab or rituximab
6. Participants who started 5-aminosalicylic acid oral drug or probiotics treatment, antimicrobials to treat Crohn's disease, or 30 mg/day or less of oral corticosteroids within 13 days before initiation of study drug administration. If these drugs were used within 14 days before initiation of study drug administration, the dosage must have been changed or their use discontinued within 13 days before the initiation of study drug administration
7. Participants who had received 5-aminosalicylic acid or corticosteroid enemas/suppositories, intravenous corticosteroid injections, or more than 30 mg/day of oral corticosteroids, medications for diarrhea-predominant irritable bowel syndrome, or Chinese herbal medicine for the treatment of Crohn's disease (e.g., Daikenchuto) within 13 days before initiation of study drug administration
8. Participants who had received azathioprine, 6-mercaptopurine, or methotrexate within 27 days before initiation of study drug administration. However, this shall not apply to participants who have received these drugs for 83 or more days before initiation of the study drug administration and continued the steady dose administration of the drugs for 27 or more days before initiation of the study drug administration
9. Participants who had received cyclosporin, tacrolimus, tofacitinib or any study drugs for treatment of ulcerative colitis within 27 days before initiation of the study drug administration
10. Participants who had received adalimumab within 27 days before initiation of study drug administration or any biological drugs other than adalimumab within 55 days before initiation of study drug administration. Topical administration (such as intraocular implantation for treatment of age-related maculopacy) is allowed
11. Participants who had received any live vaccinations within 27 days before initiation of study drug administration
12. Participants who had undergone intestinal resection within 27 days before initiation of study drug administration or those anticipated to require intestinal resection during the study
13. Participants who had received leukocytapheresis or granulocyte apheresis within 27 days before initiation of the study drug administration
14. Participants who had received intravenous hyperalimentation or total enteral nutrition within the 20 days before initiation of the study drug administration or participants who are fasted
15. Participants who had received enteral nutrition at > 900 kcal/day or started enteral nutrition at <= 900 kcal/day within the 20 days before initiation of the study drug administration. Participants receiving 900 kcal/day or less of enteral nutrition for at least 21 days before initiation of the study drug administration whom these dosage was changed or the medications were discontinued within 20 days before initiation of the study drug administration
16. Participants who had been infected with Clostridium difficile, cytomegalovirus, or any other intestinal pathogen within 27 days before the first dose of the study drug
17. Participants with evidence of adenomatous colonic polyps that need to be removed at the start of study drug administration
18. Participants with a history or an complication of dysplasia of the small or large intestine
19. Participants who were suspected to have enteritis other than CD
20. Participants who were hepatitis B surface (HBs) antigen-positive or hepatitis C virus (HCV) antibody-positive at the screening. Or participants who are hepatitis B core (HBc) antibodypositive or HBs antibody positive, even though HBs antigen-negative. However, this does not apply to participants who are only HBs antibody-positive due to hepatitis B virus (HBV) vaccination, HBV-DNA-negative, HCV antigen-negative, or HCV-RNA-negative
21. Participants who had an evidence of history of tuberculosis or a suspected history of tuberculosis (including those who have findings suggesting previous tuberculosis on chest imaging procedure at the screening). However, this does not apply to participants who had completed prophylactic isoniazid, or participants who had been receiving prophylactic isoniazid for more than 21 days before the first dose of the study drug (in the latter case, the screening period are allowed to extend up to 28 days to ensure at least 21-day prophylactic isoniazid and then the study treatment is allowed to start)
22. Participants who had positive T-SPOT test or QuantiFERON test at the screening
23. Participants who had a history or complication of identified congenital or acquire immunodeficiency syndrome (eg, not-classifiable immunodeficiency, human immunodeficiency virus [HIV] infection or organ transplantation)
24. Participants who had been affected by extraintestinal infection (eg, pneumonia, sepsis, active hepatitis or pyelonephritis) within 27 days before the first dose of the study drug
25. Participants who had a treatment history with MLN0002
26. Female participants who are lactating at the screening, or have positive urine pregnancy test either at the screening or baseline
27. Participants who had serious complications in the heart, lung, liver, kidney, metabolism, gastrointestinal system, urinary system, endocrine system or blood
28. Participants who had a history of a surgery requiring general anesthesia within 27 days before the first dose of the study drug, or with a schedule of a surgery requiring hospitalization during the study period
29. Participants who had a complication or a history of malignancy. However, this does not apply to the following participants:

    * Participants who had a curative resection of localized skin basal cell carcinoma or have completed curative radiotherapy
    * Participants who had not experienced recurrence for more than 1 year since completion of a curative resection or curative radiotherapy for skin squamous cell carcinoma
    * Participants who had not experienced recurrence for more than 3 years since completion of a curative resection or curative radiotherapy for intraepithelial carcinoma of uterine cervix For participants who had a substantially distant history of malignancy (eg, 10 years or longer without recurrence since treatment completion), the investigator and the sponsor had a discussion to decide eligibility on the basis of type of malignancy and treatment applied
30. Participants who had a history or a complication of the central nervous disorder, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
31. Participants who had any subjective symptoms in the subjective PML checklist at the screening or baseline
32. Participants who had any of the following laboratory abnormalities at the screening;

    * Hemoglobin ≤8 g/dL
    * White blood cells ≤3,000/μL
    * Lymphocytes ≤500/μL
    * Platelets ≤100,000/μL or ≥1,200,000/μL
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3×upper limit of normal (ULN)
    * Alkaline phosphatase (ALP) ≥3×ULN
    * Creatinine ≥2×ULN
33. Participants who had a history or a complication of alcohol dependence or illicit drug use within one year before the first dose of the study drug
34. Participants who had a history or a complication of psychotic disorder that could obstruct compliance with the study procedures

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Clinical Science, Study Director — Takeda
Locations (56):
- Japan (56):
  - Nagoya, Aichi-ken
  - Toyota, Aichi-ken
  - Hirosaki, Aomori
  - Abiko, Chiba
  - Kashiwa, Chiba
  - Sakura, Chiba
  - Matsuyama, Ehime
  - Chikushino-shi, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Takasaki, Gunma
  - Fukuyama, Hiroshima
  - Hatsukaichi, Hiroshima
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai, Hokkaido
  - Akashi, Hyōgo
  - Nishinomiya, Hyōgo
  - Takamatsu, Kagawa-ken
  - Kamakura, Kanagawa
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Sendai, Miyagi
  - Kurashiki, Okayama-ken
  - Moriguchi, Osaka
  - Suita, Osaka
  - Tokorozawa, Saitama
  - Ōtsu, Shiga
  - Hamamatsu, Shizuoka
  - Shimotsuke, Tochigi
  - Adachi-ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Minato-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Shūnan, Yamaguchi
  - Kofu, Yamanashi
  - Chiba
  - Fukui
  - Fukuoka
  - Hiroshima
  - Kagoshima
  - Kumamoto
  - Kyoto
  - Nagasaki
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Okamoto H, Dirks NL, Rosario M, Hori T, Hibi T. Population pharmacokinetics of vedolizumab in Asian and non-Asian patients with ulcerative colitis and Crohn's disease. Intest Res. 2021 Jan;19(1):95-105. doi: 10.5217/ir.2019.09167. Epub 2020 Jul 10. PMID 32635680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 77 investigative sites in Japan from 28 Jan 2014 to 21 May 2019.
Pre-assignment Details: Participants with moderate to severe Crohn's disease were enrolled. 157 participants enrolled in induction phase, 41 participants entered maintenance phase and 134 participants entered open-label cohort and received placebo or vedolizumab 300 mg. Open-label cohort occurred between Week 10 and 154 through study with maximum of 94 weeks of treatment.
Period: Induction Phase (Week 0 to 14)
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
Started | 79 | 78 | 0 | 0 | 0 | 0
Completed | 73 | 66 | 0 | 0 | 0 | 0
Not Completed | 6 | 12 | 0 | 0 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 3 | 11 | 0 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Phase (Week 14 to 60)
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
Started (Participants who achieved clinical response at Week 10 entered into the maintenance phase.) | 0 | 0 | 12 | 12 | 17 | 0
Completed | 0 | 0 | 7 | 4 | 5 | 0
Not Completed | 0 | 0 | 5 | 8 | 12 | 0
Not completed — Pretreatment Event/Adverse Event | 0 | 0 | 2 | 4 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 4 | 10 | 0
Period: Open Label Cohort (Week 10 to 154)
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
Started (23 out of 157 participants from induction/maintenance phase did not enter the open-label cohort.) | 0 | 0 | 0 | 0 | 0 | 134
Completed | 0 | 0 | 0 | 0 | 0 | 57
Not Completed | 0 | 0 | 0 | 0 | 0 | 77
Not completed — Pretreatment Event/Adverse Event | 0 | 0 | 0 | 0 | 0 | 43
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 23
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who entered in the induction phase.
Groups:
- Induction Phase: Vedolizumab, 300 mg: Vedolizumab 300 mg, IV infusion, once at Weeks 0, 2 and 6 in the induction phase.
- Total: Total of all reporting groups
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Total
Number analyzed (Participants) | 79 | 78 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.25) | 32.6 (10.93) | 33.3 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 51 | 52 | 103
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 79 | 78 | 157
Height [Mean (Standard Deviation); unit: cm] | 166.3 (8.73) | 166.4 (7.97) | 166.4 (8.33)
Weight [Mean (Standard Deviation); unit: kg] | 58.53 (14.095) | 55.03 (8.928) | 56.79 (11.906)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight(kg)/[height(m)^2]
  kg/m^2 | 21.15 (4.942) | 19.81 (2.567) | 20.48 (3.989)
Duration of Crohn's Disease [Median (Full Range); unit: years] — Duration between the first diagnosis of Crohn's disease and the start of the study was reported.
  years | 7.20 [0.3 to 27.8] | 8.35 [0.3 to 32.0] | 7.90 [0.3 to 32.0]
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/dL] | 2.234 (2.1763) | 2.848 (3.2303) | 2.539 (2.7593)
CDAI Score at Week 0 [Mean (Standard Deviation); unit: score on a scale] — CDAI is scoring system for the Assessment of Crohn's Disease Activity. The total CDAI score ranges from 0 to approximately 600 , where higher scores indicate more severe disease. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease.
  score on a scale | 303.9 (63.19) | 295.0 (64.81) | 299.5 (63.95)
Disease Localization [Count of Participants; unit: Participants]
  Small Intestine Type | 13 | 9 | 22
  Large Intestine Type | 11 | 19 | 30
  Small/large Intestine Type | 55 | 50 | 105
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 46 | 42 | 88
  Current Smoker | 13 | 11 | 24
  Ex-smoker | 20 | 25 | 45
Extraintestinal Manifestations (Based on CDAI subscore) [Count of Participants; unit: Participants] — CDAI is scoring system for the Assessment of Crohn's Disease Activity. The total CDAI score ranges from 0 to approximately 600, where higher scores indicate more severe disease. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease.
  Participants
    Had No Extraintestinal Manifestations | 24 | 22 | 46
    Had Extraintestinal Manifestations | 55 | 56 | 111
Extraintestinal Manifestations (Based on Case Report Form) [Count of Participants; unit: Participants]
  Had No Extraintestinal Manifestations | 42 | 52 | 94
  Had Extraintestinal Manifestations | 37 | 26 | 63
History of Prior Surgery for Crohn's Disease (CD) [Count of Participants; unit: Participants]
  Had No Surgical History | 55 | 48 | 103
  Had Surgical History | 24 | 30 | 54
Current Medical Condition Related to Fistula [Count of Participants; unit: Participants]
  Had No Current Medical Condition | 72 | 66 | 138
  Had Current Medical Condition | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Induction Phase: Percentage of Participants With Crohn's Disease Activity Index (CDAI)-100 Response
Description: A response to therapy is considered a decrease from baseline of at least 100 points in the CDAI score at Week 10. CDAI is scoring system for the assessment of Crohn's disease activity. The total CDAI score ranges from 0 to approximately 600, where higher scores indicate more severe disease. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease.
Time Frame: Week 10
Population: Full analysis set (FAS) in the induction phase included participants who were randomized and received at least one dose of the study drug in induction phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo
Number analyzed (Participants) | 79 | 78
percentage of participants | 26.6 [17.268 to 37.720] | 16.7 [9.184 to 26.813]
Statistical Analysis 1: Comparison: Induction Phase: Vedolizumab, 300 mg vs Induction Phase: Placebo; Test type: Superiority; p = 0.1448, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.816 to 3.958] — MLN0002 group/placebo group. Cochran-Mantel-Haenszel (CMH) test was used for analysis. Prior tumor necrosis factor alpha (TNFα) antagonist use (yes/no) was used as stratification factor

2. Primary Outcome: Maintenance Phase: Percentage of Participants With Clinical Remission
Description: Clinical remission is defined as the CDAI score ≤150. CDAI is scoring system for the assessment of Crohn's disease activity. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease.
Time Frame: Week 60
Population: FAS in the maintenance phase included participants who were randomized and received at least one dose of the study drug in the maintenance phase. The FAS in the maintenance phase does not include participants who received placebo in the induction phase and were enrolled into the maintenance phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maintenance Phase: Vedolizumab 300 mg: Vedolizumab placebo-matching, IV infusion, once at Weeks 14, 22, 30, 38, 46 and 54 in maintenance phase. Participants received vedolizumab in induction phase and achieved CDAI -70 response at Week 10 and were randomized to receive vedolizumab in maintenance phase.
Arm/Group | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 12 | 12
percentage of participants | 41.7 [15.165 to 72.333] | 16.7 [2.086 to 48.414]
Statistical Analysis 1: Comparison: Maintenance Phase: Vedolizumab 300 mg vs Maintenance Phase: Placebo; Test type: Superiority; p = 0.1779, Pearson's Chi-square Test; Odds Ratio (OR) = 3.57, 95% CI 2-sided [0.532 to 23.953] — MLN0002 group/placebo group

3. Primary Outcome: Number of Participants Who Experienced at Least One or More Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) is defined as any untoward medical occurrence in a study participant who received a drug (including a study drug); it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From Baseline up to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: Safety analysis set included participants who received at least one dose of the study drug in either the induction phase, the maintenance phase or the open-label cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
Number analyzed (Participants) | 79 | 78 | 12 | 12 | 17 | 134
Participants | 49 | 42 | 9 | 10 | 12 | 130

4. Primary Outcome: Number of Participants With TEAE Related to Body Weight (Weight Decreased)
Description: Reported events on this outcome measure were "Weight Decreased".
Time Frame: From Baseline up to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
Number analyzed (Participants) | 79 | 78 | 12 | 12 | 17 | 134
Participants | 0 | 0 | 0 | 0 | 0 | 2

5. Primary Outcome: Number of Participants With TEAE Related to Vital Signs
Description: Vital signs included body temperature (axilla), sitting blood pressure (after the participant has rested for at least 5 minutes), and pulse (bpm). Reported events on this outcome measure were "Pyrexia", "Body temperature increased", "Hypertension", and "Orthostatic hypotension".
Time Frame: From Baseline up to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
Number analyzed (Participants) | 79 | 78 | 12 | 12 | 17 | 134
Participants
  Pyrexia | 3 | 1 | 0 | 1 | 1 | 19
  Body Temperature Increased | 1 | 0 | 0 | 0 | 0 | 0
  Hypertension | 0 | 0 | 1 | 0 | 0 | 1
  Orthostatic Hypotension | 0 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Participants With TEAE Related to Electrocardiogram (ECG) [Bundle Branch Block Right]
Description: Reported events on this outcome measure were "Bundle Branch Block Right".
Time Frame: From Baseline up to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
Number analyzed (Participants) | 79 | 78 | 12 | 12 | 17 | 134
Participants | 0 | 0 | 0 | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Markedly Abnormal Values of Laboratory Parameters Values
Description: The laboratory values outside the range (Hemoglobin <=7 g/dL, Lymphocytes <500 /microL, White Blood Cell (WBC) <2000 /microL, Platelets <7.5 10^4/microL, Neutrophils <1000 /microL, Alanine Aminotransferase (ALT) (Glutamic Pyruvic Transaminase; GPT) >3.0 U/L x upper limit of normal (ULN), Aspartate Aminotransferase (AST) (Glutamic Oxaloacetic Transaminase; GOT) >3.0 U/L x ULN, Total Bilirubin >2.0 mg/dL x ULN, Amylase >2.0 (U/L) x ULN are considered markedly abnormal.
Time Frame: From Baseline up to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
Number analyzed (Participants) | 79 | 78 | 11 | 12 | 17 | 134
Participants
  Hemoglobin (g/dL) <=7 | 0 | 1 | 0 | 0 | 0 | 4
  Lymphocytes (/uL) <500 | 7 | 6 | 1 | 2 | 1 | 18
  WBC (/uL) <2000 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets (10^4/uL) <7.5 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophils (/uL) <1000 | 0 | 0 | 0 | 0 | 0 | 1
  ALT (GPT) (U/L) >3.0 x ULN | 1 | 1 | 0 | 0 | 0 | 1
  AST (GOT) (U/L) >3.0 x ULN | 1 | 0 | 0 | 0 | 0 | 1
  Total Bilirubin (mg/dL) >2.0 x ULN | 0 | 0 | 0 | 0 | 0 | 4
  Amylase (U/L) >2.0 x ULN | 1 | 0 | 0 | 0 | 0 | 8

8. Secondary Outcome: Induction Phase: Percentage of Participants With Clinical Remission
Description: as for outcome 2
Time Frame: Week 10
Population: FAS in the induction phase included participants who were randomized and received at least one dose of the study drug in induction phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo
Number analyzed (Participants) | 79 | 78
percentage of participants | 17.7 [10.041 to 27.942] | 10.3 [4.533 to 19.213]
Statistical Analysis 1: Comparison: Induction Phase: Vedolizumab, 300 mg vs Induction Phase: Placebo; Test type: Superiority; p = 0.1963, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.720 to 4.673] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Induction Phase: Change From Baseline in C-reactive Protein (CRP) Values
Time Frame: Baseline to Week 10
Population: Participants from 'FAS in the induction phase' with CRP value exceeding 0.30 mg/dL at Baseline were analyzed at given time point. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo
Number analyzed (Participants) | 79 | 78
mg/dL
  Change from Baseline at Week 2: number analyzed (Participants) | 64 | 70
  Change from Baseline at Week 2 | 0.022 (2.1421) | -0.125 (2.8417)
  Change from Baseline at Week 6: number analyzed (Participants) | 61 | 65
  Change from Baseline at Week 6 | -0.089 (2.0266) | 0.130 (2.1674)
  Change from Baseline at Week 10: number analyzed (Participants) | 60 | 59
  Change from Baseline at Week 10 | -0.164 (2.2729) | 0.077 (2.8690)

10. Secondary Outcome: Maintenance Phase: Percentage of Participants With Crohn's Disease Activity Index (CDAI)-100 Response
Description: as for outcome 1
Time Frame: Week 60
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 12 | 12
percentage of participants | 58.3 [27.667 to 84.835] | 8.3 [0.211 to 38.480]
Statistical Analysis 1: Comparison: Maintenance Phase: Vedolizumab 300 mg vs Maintenance Phase: Placebo; Test type: Superiority; p = 0.0094, Pearson's Chi-square Test; Odds Ratio (OR) = 15.40, 95% CI 2-sided [1.473 to 160.972]

11. Secondary Outcome: Maintenance Phase: Percentage of Participants With Durable Clinical Remission
Description: Durable clinical remission is defined as participants with CDAI score ≤ 150 at both Weeks 14 and 60. CDAI is scoring system for the assessment of Crohn's disease activity. The total CDAI score ranges from 0 to approximately 600, where higher scores indicate more severe disease. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease.
Time Frame: From Week 14 and Week 60
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 12 | 12
percentage of participants | 33.3 [9.925 to 65.112] | 25.0 [5.486 to 57.186]
Statistical Analysis 1: Comparison: Maintenance Phase: Vedolizumab 300 mg vs Maintenance Phase: Placebo; Test type: Superiority; p = 0.6534, Pearson's Chi-square Test; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.254 to 8.844] — MLN0002 group/placebo group

12. Secondary Outcome: Maintenance Phase: Percentage of Participants With Corticosteroid-free Clinical Remission
Description: Corticosteroid-free clinical remission is defined as participants using oral corticosteroids at baseline (Week 0) who discontinued corticosteroids and were in clinical remission (CDAI score ≤ 150) at Week 60. CDAI is scoring system for the assessment of Crohn's disease activity. The total CDAI score ranges from 0 to approximately 600, where higher scores indicate more severe disease. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease.
Time Frame: Week 60
Population: Participants from FAS in maintenance phase included participants who were randomized and received at least one dose of the study drug in the maintenance phase and administered oral corticosteroids concomitantly at Week 0, were analyzed at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 5 | 3
percentage of participants | 40.0 [5.274 to 85.337] | 0.0 [0.000 to 70.760]
Statistical Analysis 1: Comparison: Maintenance Phase: Vedolizumab 300 mg vs Maintenance Phase: Placebo; Test type: Superiority; p = 0.2059, Pearson's Chi-square Test

13. Secondary Outcome: Serum Vedolizumab Concentration in Induction Phase
Time Frame: Weeks 2, 6, 10 and 14
Population: Participants from 'FAS in Induction Phase', who were randomized and received at least one dose of the study drug in the induction phase and for whom samples were available for pharmacokinetic (PK) analysis. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Induction Phase: Vedolizumab, 300 mg
Number analyzed (Participants) | 79
ug/mL
  Week 2: number analyzed (Participants) | 57
  Week 2 | 28.23 (11.018)
  Week 6: number analyzed (Participants) | 50
  Week 6 | 21.01 (14.076)
  Week 10: number analyzed (Participants) | 60
  Week 10 | 22.31 (14.049)
  Week 14: number analyzed (Participants) | 17
  Week 14 | 12.24 (10.350)

14. Secondary Outcome: Serum Vedolizumab Concentration in Maintenance Phase
Time Frame: Weeks 2, 6, 10, 14, 22, 30 and 60
Population: Participants from 'FAS in Maintenance Phase', who were randomized and received at least one dose of the study drug in the maintenance phase and for whom samples were available for PK analysis. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 12 | 12
ug/mL
  Week 2: number analyzed (Participants) | 10 | 9
  Week 2 | 29.32 (13.880) | 30.54 (9.7495)
  Week 6: number analyzed (Participants) | 10 | 9
  Week 6 | 25.19 (17.054) | 24.90 (14.490)
  Week 10: number analyzed (Participants) | 11 | 9
  Week 10 | 26.24 (15.464) | 26.60 (15.642)
  Week 14: number analyzed (Participants) | 10 | 7
  Week 14 | 11.20 (8.5793) | 13.72 (13.072)
  Week 22: number analyzed (Participants) | 9 | 7
  Week 22 | 9.102 (6.1809) | 1.502 (2.8285)
  Week 30: number analyzed (Participants) | 8 | 4
  Week 30 | 9.013 (6.8774) | 0.000 (0.0000)
  Week 60: number analyzed (Participants) | 6 | 3
  Week 60 | 13.68 (4.2659) | 0.000 (0.0000)

15. Secondary Outcome: Number of Participants With Anti-vedolizumab Antibodies (AVA) in Induction Phase
Time Frame: Weeks 0, 10 and 16 weeks after the last dose of study drug in induction phase
Population: Participants who underwent proper AVA test out of 'the FAS in the induction phase' were analyzed in this outcome measure. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg
Number analyzed (Participants) | 79
Participants
  Week 0: number analyzed (Participants) | 63
  Week 0 | 1
  Week 10: number analyzed (Participants) | 63
  Week 10 | 1
  16 Weeks After Last Administration: number analyzed (Participants) | 4
  16 Weeks After Last Administration | 0

16. Secondary Outcome: Number of Participants With Anti-vedolizumab Antibodies (AVA) in Maintenance Phase
Time Frame: Weeks 0, 10, 30, 60 and 16 weeks after the last dose of study drug in maintenance phase
Population: Participants who underwent proper AVA test out of the 'FAS in Maintenance Phase', the participants who received at least one dose of study drug in the maintenance phase were analyzed in this outcome measure. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Week 0: number analyzed (Participants) | 11 | 9
  Week 0 | 0 | 0
  Week 10: number analyzed (Participants) | 11 | 9
  Week 10 | 0 | 0
  Week 30: number analyzed (Participants) | 10 | 9
  Week 30 | 0 | 2
  Week 60: number analyzed (Participants) | 9 | 4
  Week 60 | 0 | 1
  16 Weeks After Last Administration: number analyzed (Participants) | 1 | 1
  16 Weeks After Last Administration | 0 | 0

17. Secondary Outcome: Number of Participants With Anti-vedolizumab Antibodies (AVA) in Open Label Cohort
Time Frame: Weeks 0, 10, 30, 62, 94 and 16 weeks after the last dose of study drug in open-label cohort
Population: Participants who underwent proper AVA test out of the 'FAS in Open Label Cohort', the participants who received at least one dose of study drug in the open label cohort were analyzed in this outcome measure. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label: Vedolizumab 300 mg
Number analyzed (Participants) | 134
Participants
  Week 0: number analyzed (Participants) | 57
  Week 0 | 2
  Week 10: number analyzed (Participants) | 108
  Week 10 | 2
  Week 30: number analyzed (Participants) | 94
  Week 30 | 2
  Week 62: number analyzed (Participants) | 66
  Week 62 | 0
  Week 94: number analyzed (Participants) | 49
  Week 94 | 0
  16 Weeks After Last Administration: number analyzed (Participants) | 98
  16 Weeks After Last Administration | 2

18. Secondary Outcome: Number of Participants With Neutralizing Anti-vedolizumab Antibodies (AVA) in Induction Phase
Time Frame: Weeks 0, 10 and 16 weeks after the last dose of study drug in induction phase
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Vedolizumab, 300 mg
Number analyzed (Participants) | 79
Participants
  Week 0: number analyzed (Participants) | 63
  Week 0 | 0
  Week 10: number analyzed (Participants) | 63
  Week 10 | 1
  16 Weeks After Last Administration: number analyzed (Participants) | 4
  16 Weeks After Last Administration | 0

19. Secondary Outcome: Number of Participants With Neutralizing Anti-vedolizumab Antibodies (AVA) in Maintenance Phase
Time Frame: Weeks 0, 10, 30, 60 and 16 weeks after the last dose of study drug in maintenance phase
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Week 0: number analyzed (Participants) | 11 | 9
  Week 0 | 0 | 0
  Week 10: number analyzed (Participants) | 11 | 9
  Week 10 | 0 | 0
  Week 30: number analyzed (Participants) | 10 | 9
  Week 30 | 0 | 2
  Week 60: number analyzed (Participants) | 9 | 4
  Week 60 | 0 | 1
  16 Weeks After Last Administration: number analyzed (Participants) | 1 | 1
  16 Weeks After Last Administration | 0 | 0

20. Secondary Outcome: Number of Participants With Neutralizing Anti-vedolizumab Antibodies (AVA) in Open Label Cohort
Time Frame: Weeks 0, 10, 30, 62, 94 and 16 weeks after the last dose of study drug in open-label cohort
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label: Vedolizumab 300 mg
Number analyzed (Participants) | 134
Participants
  Week 0: number analyzed (Participants) | 57
  Week 0 | 2
  Week 10: number analyzed (Participants) | 108
  Week 10 | 2
  Week 30: number analyzed (Participants) | 94
  Week 30 | 1
  Week 62: number analyzed (Participants) | 66
  Week 62 | 0
  Week 94: number analyzed (Participants) | 49
  Week 94 | 0
  16 Weeks After Last Administration: number analyzed (Participants) | 98
  16 Weeks After Last Administration | 2

ADVERSE EVENTS:
Time Frame: From Baseline up to 16 weeks after the last dose of study drug (Up to approximately 170 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Induction Phase: Vedolizumab, 300 mg | Induction Phase: Placebo | Maintenance Phase: Vedolizumab 300 mg | Maintenance Phase: Placebo | Maintenance Phase: Placebo Continuation | Open-Label: Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/78 | 0/12 | 0/12 | 0/17 | 0/134
Serious Adverse Events (participants affected / at risk) | 8/79 | 10/78 | 2/12 | 4/12 | 2/17 | 70/134
Other Adverse Events (participants affected / at risk) | 17/79 | 19/78 | 9/12 | 7/12 | 12/17 | 113/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Vedolizumab, 300 mg (N=79) | Induction Phase: Placebo (N=78) | Maintenance Phase: Vedolizumab 300 mg (N=12) | Maintenance Phase: Placebo (N=12) | Maintenance Phase: Placebo Continuation (N=17) | Open-Label: Vedolizumab 300 mg (N=134)
Crohn's disease (Gastrointestinal disorders) | 2 | 10 | 1 | 2 | 1 | 35
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 4
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anaphylactoid reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Mesenteric abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Mycotic endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Periumbilical abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyslalia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intracranial hypotension (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Vedolizumab, 300 mg (N=79) | Induction Phase: Placebo (N=78) | Maintenance Phase: Vedolizumab 300 mg (N=12) | Maintenance Phase: Placebo (N=12) | Maintenance Phase: Placebo Continuation (N=17) | Open-Label: Vedolizumab 300 mg (N=134)
Crohn's disease (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 2 | 27
Nasopharyngitis (Infections and infestations) | 11 | 11 | 4 | 4 | 4 | 55
Enteritis infectious (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 0 | 0 | 0 | 9
Hypoaesthesia (Nervous system disorders) | 4 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 9
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 15
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 11
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 19
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Allergy to metals (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 10
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 13
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 10
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 16
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 8
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 8
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2013-11-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT02038920/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT02038920/SAP_001.pdf